CLINICAL TRIAL: NCT01010750
Title: A Phase I, Randomized, Double Blind, Three-Period Crossover, Estimation Study Using Lisdexamfetamine Dimesylate, Immediate Release Mixed Amphetamine Salts and Placebo to Evaluate the Utility of a Standardized Computer Battery of Tests in Adults With Attention-Deficit Hyperactivity Disorder (ADHD)
Brief Title: Lisdexamfetamine Dimesylate (LDX) Pilot Cognition Study to Evaluate the Utility of a Standardized Battery of Tests in Adults With Attention-Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: SPD489-115
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Attention-Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- LDX + MAS-IR Placebo (Active Comparator): Lisdexamfetamine Dimesylate (LDX) + Immediate Release Mixed Amphetamine Salts (MAS-IR) placebo
  Interventions: Drug: Lisdexamfetamine Dimesylate (LDX)
- MAS-IR + LDX Placebo (Active Comparator): Immediate Release Mixed Amphetamine Salts (MAS-IR) + Lisdexamfetamine Dimesylate (LDX) placebo
  Interventions: Drug: Immediate Release Mixed Amphetamine Salts (MAS-IR)
- Placebo (Placebo Comparator): Lisdexamfetamine Dimesylate (LDX) Placebo + Immediate Release Mixed Amphetamine Salts (MAS-IR) Placebo
  Interventions: Drug: LDX Placebo + MAS-IR Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate (LDX) — Lisdexamfetamine Dimesylate (LDX) + Immediate Release Mixed Amphetamine Salts (MAS-IR) placebo
  Arms: LDX + MAS-IR Placebo
Drug: Immediate Release Mixed Amphetamine Salts (MAS-IR) — Immediate Release Mixed Amphetamine Salts (MAS-IR) + Lisdexamfetamine Dimesylate (LDX) placebo
  Arms: MAS-IR + LDX Placebo
Drug: LDX Placebo + MAS-IR Placebo — Lisdexamfetamine Dimesylate (LDX) Placebo + Immediate Release Mixed Amphetamine Salts (MAS-IR) Placebo
  Arms: Placebo

SUMMARY:
To evaluate the sensitivity and responsiveness of a standardized, validated, computer-based, battery of neuro-psychometric tests in adults with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Subject meets Diagnostic and Statistical Manual of Mental Disorders Fourth Edition; Text Revision (DSM IV TR) criteria for a primary diagnosis of ADHD (diagnostic code 314.00 and 314.01) established by a comprehensive psychiatric evaluation that reviews DSM-IV-TR criteria with at least 6 of the 9 subtype criteria met.
2. Subject has been previously treated for ADHD with an adequate course of amphetamine therapy with no history of intolerance, or lack of efficacy, as determined by the Investigator.
3. Subject does not have any physical disability (eg. colorblindness, limitations with use of one or both hands, etc) that would interfere with the subject's participation in or performance on any of the neuropsychometric tests. For a number of these tasks speed is a key factor thus subjects cannot have any obvious impediments/impairments in the use of their hands.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01-05 (Actual); Primary Completion 2010-03-28 (Actual); Study Completion 2010-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Claghorn-Lesem Research Clinic, Houston, Texas, United States

REFERENCES:
- [Result] Martin PT, Corcoran M, Zhang P, Katic A. Randomized, double-blind, placebo-controlled, crossover study of the effects of lisdexamfetamine dimesylate and mixed amphetamine salts on cognition throughout the day in adults with attention-deficit/hyperactivity disorder. Clin Drug Investig. 2014 Feb;34(2):147-57. doi: 10.1007/s40261-013-0156-z. PMID 24297663
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each of the 3 treatment regimens was administered daily for 7 days (a total of 21 days of treatment). There was no washout between regimens.
Groups:
- LDX 50 mg First, Then MAS-IR 20 mg, Then Placebo: Lisdexamfetamine Dimesylate (LDX) 50 mg + Immediate Release Mixed Amphetamine Salts (MAS-IR) placebo first, then MAS-IR 20 mg + LDX placebo, then LDX placebo + MAS-IR placebo
- LDX 50 mg First, Then Placebo, Then MAS-IR 20 mg: LDX 50 mg + MAS-IR placebo first, then LDX placebo + MAS-IR placebo, then MAS-IR 20 mg + LDX placebo
- Placebo First, Then LDX 50 mg, Then MAS-IR 20 mg: LDX placebo + MAS-IR placebo first, then LDX 50 mg + MAS-IR placebo, then MAS-IR 20 mg + LDX placebo
- Placebo First, Then MAS-IR 20 mg, Then LDX 50 mg: LDX placebo + MAS-IR placebo first, then MAS-IR 20 mg + LDX placebo, then LDX 50 mg + MAS-IR placebo
- MAS-IR 20 mg First, Then LDX 50 mg, Then Placebo: MAS-IR 20 mg + LDX placebo first, then LDX 50 mg + MAS-IR placebo, then LDX placebo + MAS-IR placebo
- MAS-IR 20 mg First, Then Placebo, Then LDX 50 mg: MAS-IR 20 mg + LDX placebo first, then LDX placebo + MAS-IR placebo, then LDX 50 mg + MAS-IR placebo
Period: First Intervention
Arm/Group | LDX 50 mg First, Then MAS-IR 20 mg, Then Placebo | LDX 50 mg First, Then Placebo, Then MAS-IR 20 mg | Placebo First, Then LDX 50 mg, Then MAS-IR 20 mg | Placebo First, Then MAS-IR 20 mg, Then LDX 50 mg | MAS-IR 20 mg First, Then LDX 50 mg, Then Placebo | MAS-IR 20 mg First, Then Placebo, Then LDX 50 mg
Started | 3 | 4 | 3 | 3 | 2 | 3
Completed | 3 | 4 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | LDX 50 mg First, Then MAS-IR 20 mg, Then Placebo | LDX 50 mg First, Then Placebo, Then MAS-IR 20 mg | Placebo First, Then LDX 50 mg, Then MAS-IR 20 mg | Placebo First, Then MAS-IR 20 mg, Then LDX 50 mg | MAS-IR 20 mg First, Then LDX 50 mg, Then Placebo | MAS-IR 20 mg First, Then Placebo, Then LDX 50 mg
Started | 3 | 4 | 3 | 3 | 2 | 3
Completed | 3 | 3 | 3 | 3 | 2 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | LDX 50 mg First, Then MAS-IR 20 mg, Then Placebo | LDX 50 mg First, Then Placebo, Then MAS-IR 20 mg | Placebo First, Then LDX 50 mg, Then MAS-IR 20 mg | Placebo First, Then MAS-IR 20 mg, Then LDX 50 mg | MAS-IR 20 mg First, Then LDX 50 mg, Then Placebo | MAS-IR 20 mg First, Then Placebo, Then LDX 50 mg
Started | 3 | 3 | 3 | 3 | 2 | 3
Completed | 3 | 3 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LDX 50 mg First, Then MAS-IR 20 mg, Then Placebo | LDX 50 mg First, Then Placebo, Then MAS-IR 20 mg | Placebo First, Them LDX 50 mg, Then MAS-IR 20 mg | Placebo First, Then MAS-IR 20 mg, Then LDX 50 mg | MAS-IR 20 mg First, Then LDX 50 mg, Then Placebo | MAS-IR 20 mg First, Then Placebo, Then LDX 50 mg | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 2 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (1.00) | 24.8 (6.70) | 30.3 (6.11) | 31.3 (11.37) | 53.0 (0.00) | 30.0 (11.36) | 30.8 (10.75)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 55 years | 3 | 4 | 3 | 3 | 2 | 3 | 18
  >=56 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 1 | 1 | 2 | 7
  Male | 3 | 2 | 2 | 2 | 1 | 1 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 4 | 3 | 3 | 2 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Power of Attention Score
Description: The Power of Attention score reflects the ability to focus attention, and is calculated as the sum of the reaction time, measured in milliseconds, from 3 attention tests (Simple Reaction Time, Choice Reaction Time, and Digit Vigilance Speed). Faster performance (lower times) reflects more intense concentration. A decrease in the Power of Attention score indicates improvement.
Time Frame: pre-dose and at 1, 2, 3, 4, 5, 8, 12, 14 and 16 hours post-dose on Day 7
Population: The Pharmacodynamic Set (PD) is all subjects in the Safety Set who had at least 1 post-dose assessment of the pharmacodynamic variables. The Safety Set contains all enrolled subjects who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | LDX 50 mg | MAS-IR 20 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 17
milliseconds
  half an hour prior to dosing | 1260.7 (34.000) | 1324.1 (47.142) | 1272.8 (33.729)
  1 hour post-dose | 1244.6 (32.887) | 1307.4 (42.908) | 1253.1 (24.174)
  2 hours post-dose | 1315.5 (67.246) | 1255.0 (33.905) | 1296.2 (39.808)
  3 hours post-dose | 1219.1 (33.428) | 1229.6 (37.865) | 1301.0 (40.864)
  4 hours post-dose | 1225.9 (40.192) | 1236.5 (36.839) | 1275.4 (35.302)
  5 hours post-dose | 1179.6 (35.022) | 1251.4 (42.607) | 1330.3 (49.623)
  8 hours post-dose | 1212.0 (36.113) | 1259.3 (35.883) | 1304.5 (43.802)
  12 hours post-dose | 1232.4 (48.183) | 1239.3 (38.465) | 1262.1 (40.795)
  14 hours post-dose | 1199.3 (35.947) | 1270.1 (39.539) | 1270.5 (44.814)
  16 hours post-dose | 1202.6 (37.135) | 1255.9 (36.378) | 1270.3 (48.581)

2. Secondary Outcome: Conners Adult ADHD Rating Scales-Self Report: Short Version (CAARS-S:S) Subscale Total Score (T-Score): Inattention/Memory Problems
Description: Consists of 5 items with each item rated on a scale of 0-3 (not at all, just a little, pretty much, very much). The T-score is then calculated as: T = 50 + 10 * (raw score - mean)/Standard Deviation. The average score is 50. Scores below 50 are better than scores above 50.
Time Frame: 2 and 14 hours post-dose on Day 7
Population: PD
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LDX 50 mg | MAS-IR 20 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 17
Units on a scale
  2 hours post-dose | 66.16 (2.927) | 63.39 (3.319) | 64.92 (2.775)
  14 hours post-dose | 65.78 (3.029) | 64.45 (2.483) | 66.33 (2.398)

3. Secondary Outcome: CAARS-S:S Subscale T-Score: Hyperactivity/Restlessness
Description: as for outcome 2
Time Frame: 2 and 14 hours post-dose on Day 7
Population: PD
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LDX 50 mg | MAS-IR 20 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 17
Units on a scale
  2 hours post-dose | 64.21 (2.996) | 63.62 (3.372) | 63.28 (3.063)
  14 hours post-dose | 65.08 (2.837) | 63.41 (2.763) | 65.74 (2.597)

4. Secondary Outcome: CAARS-S:S Subscale T-Score: Impulsivity/Emotional Liability
Description: as for outcome 2
Time Frame: 2 and 14 hours post-dose on Day 7
Population: PD
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LDX 50 mg | MAS-IR 20 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 17
Units on a scale
  2 hours post-dose | 55.46 (2.931) | 54.58 (3.470) | 54.66 (3.421)
  14 hours post-dose | 57.82 (3.479) | 51.53 (2.802) | 55.78 (2.773)

5. Secondary Outcome: CAARS-S:S Subscale T-Score: Problems With Self-Concept
Description: as for outcome 2
Time Frame: 2 and 14 hours post-dose on Day 7
Population: PD
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LDX 50 mg | MAS-IR 20 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 17
Units on a scale
  2 hours post-dose | 58.71 (3.533) | 59.78 (3.390) | 58.40 (3.279)
  14 hours post-dose | 59.68 (3.841) | 59.54 (3.574) | 59.68 (3.055)

6. Secondary Outcome: CAARS-S:S Subscale T-Score: Attention Deficit Hyperactivity Disorder (ADHD) Index
Description: Consists of 12 items with each item rated on a scale of 0-3 (not at all, just a little, pretty much, very much). The T-score is then calculated as: T = 50 + 10 * (raw score - mean)/Standard Deviation. The average score is 50. Scores below 50 are better than scores above 50.
Time Frame: 2 and 14 hours post-dose on Day 7
Population: PD
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LDX 50 mg | MAS-IR 20 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 17
Units on a scale
  2 hours post-dose | 64.82 (3.147) | 63.90 (3.766) | 64.59 (3.681)
  14 hours post-dose | 66.56 (3.714) | 63.09 (2.945) | 64.85 (3.118)

ADVERSE EVENTS:
Description: Safety Set includes all enrolled subjects who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Arm/Group | LDX 50 mg | MAS-IR 20 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 12/18 | 9/17 | 8/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LDX 50 mg (N=18) | MAS-IR 20 mg (N=17) | Placebo (N=17)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Bruxism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Obsessive-Compulsive Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Micturition Disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 6 (8) | 4 (6) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling Jittery (General disorders) | 1 (1) | 2 (3) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Heart Rate Increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 3 (3) | 4 (5) | 1 (1)
Sensation of Heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.